CLINICAL TRIAL: NCT00097032
Title: Differences in Cognitive Function Due to Acute Sedative Effects of Risperidone and Quetiapine in Stable Bipolar I Out-Patients.
Brief Title: Study Measuring Differences in Cognition Due to Sedative Effects of Risperidone and Quetiapine in Stable Bipolar I Outpatients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Janssen, LP (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: CR004654; RIS-OUT-184
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2010-03

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I Disorder; risperidone; quetiapine; sedation; cognition
MeSH Terms: conditions — Bipolar Disorder | interventions — Risperidone; Quetiapine Fumarate

INTERVENTIONS:
Drug: risperidone; quetiapine

SUMMARY:
The purpose of this study is to determine whether the sedating (causing sleepiness) effects of risperidone or quetiapine alter cognitive (person's ability to think, perceive, recognize, remember, judge, and reason) functioning in subjects with stable Bipolar I Disorder.

DETAILED DESCRIPTION:
To compare the treatment effects of risperidone and quetiapine on cognitive function, using measures commonly believed to be affected by sedation and at doses typically used in clinical settings in stable bipolar I outpatients.One-half of patients are randomized to treatment sequence risperidone-quetiapine (R-Q), and the other one-half to quetiapine-risperidone (Q-R). Patients randomized to R-Q receive 2 mg of risperidone with dinner the night before testing and placebo with breakfast on the day of testing. After a 6 - 14 day washout period they receive 100 mg quetiapine with dinner the night before their second day of testing and 100 mg with breakfast the day of testing.

Those randomized to Q-R receive the same treatments, but in reverse order. Patients randomized to R-Q receive 2 mg of risperidone with dinner the night before testing and placebo with breakfast on the day of testing. After a 6-14 day washout period they receive 100 mg quetiapine with dinner the night before their second day of testing and 100 mg with breakfast the day of testing. Those randomized to Q-R receive the same treatments, but in reverse order.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with bipolar I disorder in partial or full remission and deemed clinically stable

Exclusion Criteria:

* Current use of benzodiazepines, prescription or herbal sleep agents
* Use of antihistamines
* Use of antipsychotic medications in the past 6 months
* Pregnant/breastfeeding females
* Females not using contraception
* Illicit drug users

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2004-10; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
To compare the treatment effects of risperidone and quetiapine on cognitive function due to sedation

SECONDARY OUTCOMES:
To assess the association between subjective experience of sedation and cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Harvey PD, Hassman H, Mao L, Gharabawi GM, Mahmoud RA, Engelhart LM. Cognitive functioning and acute sedative effects of risperidone and quetiapine in patients with stable bipolar I disorder: a randomized, double-blind, crossover study. J Clin Psychiatry. 2007 Aug;68(8):1186-94. doi: 10.4088/jcp.v68n0804. PMID 17854242
- See also: Study Measuring Differences in Cognition Due to Sedative Effects of Risperidone and Quetiapine in Stable Bipolar I Outpatients — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1086&filename=CR004654_CSR.pdf